CLINICAL TRIAL: NCT00664339
Title: Influenza Vaccine Pilot Study in Severe Congestive Heart Failure Patients. The Flu Vaccination Heart Failure (FLUVACS II) Study
Brief Title: Flu Vaccination in Congestive Heart Failure
Acronym: FLUVACS-IC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: La Fundacion Favaloro para la Investigacion y la Docencia Medica (Other)
Responsible Party: ENRIQUE P. GURFINKEL, MD PhD, Fundacion Favaloro para la Docencia y la Investigacion Medica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DDI (976) 407
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Heart Failure
Keywords: Heart failure,; infection,; immune system,; atherosclerosis
MeSH Terms: conditions — Heart Failure; Infections; Atherosclerosis | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Active Comparator): Flu Vaccine
  Interventions: Biological: Flu Vaccine
- Control (Other): Conventional treatment therapy for heart failure
  Interventions: Other: Conventional medical therapy for heart failure

INTERVENTIONS:
Biological: Flu Vaccine — Single dose of Flu vaccine by year (1)
  Arms: Vaccine
Other: Conventional medical therapy for heart failure — According with the international guidelines
  Arms: Control

SUMMARY:
We evaluated the preventive impact of vaccination on subsequent death events in 117 severe congestive heart patients requiring ventilator support without endotracheal intubations and aggressive medical therapy.

They were randomly allocated in a single-blind manner as a unique intramuscular influenza vaccination or as controls.

The first primary outcome evaluated at 6 months follow-up - cardiovascular death - occurred in 3% of the patients in the vaccine group Vs 17% in controls (p=0.022). The composite end point occurred in 33% of the patients in the vaccine group Vs 74% in control group, p = <0.001.

DETAILED DESCRIPTION:
Background: Recent reports detected that one of the barriers that vaccination against influenza infection is that, physicians do not strongly recommend its applications to cardiovascular patients at risk. We evaluated the preventive impact of vaccination against death in severe congestive heart failure hospitalized patients.

Methods and Results: A total of 117 severe congestive heart failure patients (New York Heart Association class III and IV) admitted in the first 12 hours who required ventilator support without endotracheal intubations and high doses of loop-diuretics, were included in a prospective, multicenter log, during the winter season. Congestive heart patients received intravenous vasodilators and loop-diuretics plus standard therapies, and then were randomly allocated in a single-blind manner as a unique intramuscular influenza vaccination or as controls. Death, and combined end points (death, and re-hospitalization for any reason) were assessed at 6 months follow-up.

The first primary outcome - cardiovascular death - occurred in 3% of the patients in the vaccine group Vs 17% in controls (odds ratio with vaccine as compared with controls: 0.16; 95 percent confidence interval, 0.33 to 0.79; p=0.022). The composite end point occurred in 33% of the patients in the vaccine group Vs 74% in controls, p = <0.001. The need of adding inotropic drugs occurred in 8% of patients receiving vaccination, and in 12.5% in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient's > 21 years of age with a severe congestive heart failure (New York Heart Association class III or IV) requiring an immediate administration of intravenous vasodilators drugs, oxygen therapy, and no less than 160 mg of intravenous furosemide were eligible for inclusion.
* Definite evidence of underlying heart failure was also required as shown by at least two of the following:

  * a) Orthopnea on admission
  * b) X-ray showing evidences of elevated wedge pressure indicating congestive heart failure
  * c) recent prior hospitalization (within the 30 days prior to the index hospitalization) because a congestive heart failure episode
  * d) echocardiography data showing a poor left ventricular ejection fraction (0.40 or lower measuring with the biplane Simpson's method
  * e) non-invasive ventilation to the maintenance of SaO2 above 90%
  * f) wet rales in at least the lower half of the lungs fields
* Patients with a final diagnosis of Congestive Heart Failure as a consequence of necrotic or chronic ischemic heart disease, or infective origin such as chronic Chagas Disease, chronic valvular heart disease (surgically repaired or not), and idiopathic origin were also included for the present study

Exclusion Criteria:

* Patients with a concomitant infective disease were excluded from the study
* Patients with evidence of evolving with multi organic failure (hepatic or renal dysfunction requiring dialysis), terminal disease, or any impeding cause of follow-up, including contraindications of vaccination, were excluded from the study
* Those with congestive heart failure following unstable coronary artery disease, or prior by-pass surgery, or angioplasty or congestive heart failure complicating myocardial infarction requiring urgent intervention were excluded also
* Those individuals who required mechanical ventilation on admission
* Patients with prior vaccinations were also excluded
* Pregnancy condition was an exclusion criterion
* Those patients who were unable or refused to give a written inform consent was also excluded of the present study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Total Death | 6 mounths

SECONDARY OUTCOMES:
Rehospitalization for any cause or infarction | 6 mounths

CONTACTS AND LOCATIONS:
Overall Officials: ENRIQUE P GURFINKEL, MD PhD, Study Chair — FUNDACION FAVALORO PARA LA DOCENCIA Y LA INVESTIGACION MEDICA